CLINICAL TRIAL: NCT04112394
Title: Evaluation of Postoperative Pain and Recovery Quality (QoR-40) in Patients Undergoing Erector Spinal Area (ESP) Block After Laparoscopic Cholecystectomy
Brief Title: Does Erector Spinal Block Improve Quality of Recovery After Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Betul Kozanhan, Ass.Prof., Konya Meram State Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ESP-Quality of Recovery
Record Dates: First submitted 2019-09-30; First posted 2019-10-02 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Postoperative Recovery
MeSH Terms: interventions — Anesthetics, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP Group (Experimental): In addition to routine standard perioperative and postoperative analgesia protocol patients will receive a single shot of local anesthetic injection at the erector spinae plane.
  Interventions: Other: local anesthetic injection
- Control (Other): Patients will receive standard perioperative and postoperative analgesia protocol.
  Interventions: Other: Standard perioperative and postoperative analgesia protocol.

INTERVENTIONS:
Other: local anesthetic injection — A linear ultrasound transducer will be place in a longitudinal parasagittal orientation about 3 cm lateral to spinous process. Local anesthetic mixture will be injected bilaterally into the fascial plane on the deep aspect of erector spinae muscle. Standard perioperative and postoperative analgesia protocol will be given and postoperative pain levels will be determined by Numerical rating scale (NRS).
  Arms: ESP Group
Other: Standard perioperative and postoperative analgesia protocol. — Standard perioperative and postoperative analgesia protocol will be given consisting of paracetamol 1 gr IV and tenoxicam 20 mg IV initiated after induction of anesthesia. At the end of the operation patients will receive contramal 1 mg/kg IV before extubation. Postoperative pain levels will be determined by Numeric Rating Scale (NRS) system, 20 minutes intervals in the first hour and at 2th, 6th, 12th and 24 th hour. For the first hour in the postoperative care unit, tramadol 50 mg IV will be given for rescue analgesia with minimum 20 minutes between doses, in patients showing a NRS ≥ 4. Paracetamol 1 g / 12 hour will be given during ward follow-up. In the ward in patients showing a NRS ≥ 4 tramadol 50 mg IV will be given for analgesia.
  Arms: Control

SUMMARY:
The primary aim of this prospective, randomized study is to evaluate the effect of erector spinae block (ESP) on quality of recovery with the QoR-40 questionnaire in patients undergoing elective laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy, one of the most common general surgical procedures, is the gold standard for the treatment of symptomatic gallbladder diseases. Although it is considered as minimally invasive surgery, pain in the early postoperative period is still meaningful. Proper pain control is essential for optimizing clinical outcomes and earlier ambulation after surgery. Traditional pain management with opioids provide good pain control, however, have undesirable side effects such as nausea, vomiting, and respiratory depression. Multimodal analgesia strategies with different classes of analgesics or local anesthetics may enhance pain relief and reduce side effects after surgery. The ESP a newer regional nerve blockade, has been used as part of a multimodal strategy to optimize postoperative pain control. The primary aim of this study is to evaluate the effect of ESP block on postoperative recovery quality in patients undergoing laparoscopic cholecystectomy with QoR-40 recovery questionnaire. Secondary aim is to assess the effect of ESP block on postoperative pain, nausea, and vomiting.

Study hypothesize is that patients who receive an ESP block in addition to the current standard of care, consisting of parenteral opioids and paracetamol, will have a clinically significant improvement in their QoR-40 at postoperative day 1 and lower pain levels, as measured by NRS in comparison to those patients who receive the current standard of care along.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) physical status I-II
* Scheduled for elective laparoscopic cholecystectomy

Exclusion Criteria:

* a history of allergy to local anesthetics
* known coagulation disorders
* infection near the puncture site
* Chronic opioid intake
* Patient with psychiatric disorders
* inability to communicate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2019-09-29 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-04-04 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery (QoR-40) score | postoperative 24 hour
  QoR-40, a 40-item questionnaire that provides a global score and subscores across five dimensions: patient support, comfort, emotions, physical independence, and pain. Each item is rated on a scale of 1-5, providing a minimum score of 40 and maximum of 200.

SECONDARY OUTCOMES:
Postoperative pain: numeric rating scale (NRS) | Postoperative 24 hours
  NRS use numbers to rate pain from 0 (no pain) to 10 (worst pain).
Analgesic consumption | Postoperative 24 hour
  Total opioid consumption after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Canıtez, Principal Investigator — M.D.
Locations (1):
- Konya Education and Training Hospital, Konya, Turkey (Türkiye)

REFERENCES:
- [Derived] Canitez A, Kozanhan B, Aksoy N, Yildiz M, Tutar MS. Effect of erector spinae plane block on the postoperative quality of recovery after laparoscopic cholecystectomy: a prospective double-blind study. Br J Anaesth. 2021 Oct;127(4):629-635. doi: 10.1016/j.bja.2021.06.030. Epub 2021 Jul 31. PMID 34340839